CLINICAL TRIAL: NCT01808807
Title: Factors Influencing Cesarean Section Rate: Does the Audit Still Work?
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief, Department of Obstetrics & Gynecology, Far Eastern Memorial Hospital
Other Study IDs: 101110-F
Record Dates: First submitted 2012-12-11; First posted 2013-03-11 (Estimated); Last update posted 2013-08-19 (Estimated); Status verified 2013-03

CONDITIONS: Cesarean Section
Keywords: cesarean section rate; the cesarean section rate audit

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- cesarean section rate after audit: cesarean section rate after audit

SUMMARY:
To elucidate the audit's effect on caesarean section rate, and also define the factors influencing the caesarean section rate.

From Jan 2007 , pregnant women who delivered in a medical center will be included retrospectively in this study. Our monthly cesarean section audit, focusing on discussing the indications of cesarean section, began from July 2008. Clinical data, indications of cesarean section, and perinatal outcomes were compared between the cases of before and after the audit. Multivariate logistic regression was performed to identify factors affecting cesarean section rate.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women who delivered in a medical center will be included retrospectively in this study

Exclusion Criteria:

* All pregnant women who delivered in a medical center will be included retrospectively in this study , no exclusion criteria

Ages: 15 Years to 47 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: pregnant women who delivered in a medical center will be included retrospectively in this study
Sampling Method: Probability Sample
Enrollment: 4000 (Actual)
Dates: Start 2012-12; Primary Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
the impact of the cesarean section rate audit | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Far Eastern Memorial Hospital, Banqiao District, Taiwan